CLINICAL TRIAL: NCT01535105
Title: Impairment in Glucose Homeostasis Among Obese Adolescents in High Risk Diabetes Prone Population - Jisr Az-Zarqa Village
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Gl homeostasis and obesity
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2012-02

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese Adolescents

SUMMARY:
Obesity is increasing all over the world in adults, adolescents and children,and is followed by morbidity, including the metabolic syndrome.

Hypothesis: Among obese adolescents there is a subgroup with impaired glucose homeostasis

The aim of the study is to identify adolescents with impaired glucose metabolism, 12-18 years, among high risk diabetes prone population, for diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of obesity

Exclusion Criteria:

* History of disease or drug therapy affecting glucose metabolism

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects of the study will be selected from a primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of Impaired Glucose Homeostasis among obese adolescents in high risk diabetes prone population | one year

SECONDARY OUTCOMES:
Description of the metabolic profile in obese adolescents | One year

CONTACTS AND LOCATIONS:
Overall Officials: Nehama Zuckerman-Levin, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit Health Services Clinic, Jisr az-Zarqa Village, Israel